CLINICAL TRIAL: NCT04435678
Title: Diagnostic Accuracy of the MADx Multi Array Xplorer (MAX 45k) Automated Laboratory System and the MADx Allergy Explorer Version 2 (ALEX²) - IgE Multiplex Test for the Diagnosis of Pre-defined Groups of Specific High-priority Allergens
Acronym: MADMAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MacroArray Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 32-332 ex 19/20
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-02

CONDITIONS: Birch Pollen Allergy; Grass Pollen Allergy; House Dust Mite Allergy; Cat Allergy; Bee Venom Allergy; Vespid Venom Allergy
MeSH Terms: conditions — Dust Mite Allergy; Venom Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- birch pollen allergy (Other): 106 patients with suspicion of birch pollen allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and a skin prick test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- grass pollen allergy (Other): 106 patients with suspicion of grass pollen allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and a skin prick test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- house dust mite allergy (Other): 148 patients with suspicion of house dust mite allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and a skin prick test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system)
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- cat allergy (Other): 106 patients with suspicion of cat allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and a skin prick test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- bee venom allergy (Other): 106 patients with suspicion of bee venom allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and an intradermal test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- vespid venom allergy (Other): 106 patients with suspicion of vespid venom allergy will be included in the study. For routine diagnosis, blood samples will be taken to determine total IgE and specific IgE and an intradermal test will be performed.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system
- non-allergic individuals (Other): 148 non-allergic individuals will be included in the study. They should have no symptoms that could be related to inhalant allergy or Hymenoptera venom allergy, negative skin test results and undetectable IgE levels.
  Left over blood samples will be used to perform the additional allergy test (ALEX² test using the MAX 45k automated laboratory system).
  Interventions: Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system

INTERVENTIONS:
Diagnostic Test: ALEX² test using the MAX 45k automated laboratory system — The ALEX² test system is a quantitative in vitro diagnostic (IVD) test for the measurement of allergen specific IgE (sIgE) and a semi-quantitative in vitro diagnostic test for the measurement of total IgE (tIgE) in human serum or plasma (exception EDTA plasma).
  The MAX 45k analyzer is intended for an automated in-vitro diagnostics use for quantitative determination of allergen specific Immunoglobulin E and semi-quantitative determination of total IgE. The MAX 45k is suitable for human serum or plasma (Heparin, Citrat, but no EDTA). MAX 45k is intended to be used only in conjunction with RAPTOR SERVER analysis software and ALEX based technology arrays.

SUMMARY:
About 20% of the general population are affected by an allergy - with an upward trend. Quite often, allergic people do not consider their disease as serious and suffer from subsequent complications, like allergic asthma, later in their life. The sooner the allergen source is identified, the sooner the therapeutic intervention (e.g. dietary recommendations, allergen avoidance, anti-inflammatory treatment or allergen immunotherapy) can be started. Cross-reactivity may also play an important role. Therefore, a comprehensive allergy test is essential for an optimal treatment of patients.

Modern multiplex testing is an individualized diagnostic approach, which may help to identify eligible patients for allergen immunotherapy and may identify risk groups by analyzing the sIgE profile. Until now, published data on the clinical usability of multiplex allergy diagnostic test systems are often limited. Even though, available studies show a good correlation between conventionally used multiplex or singleplex assays (ISAC or ImmunoCAP) and the new multiplex assay (ALEX and ALEX²), the results are often based on small sample sizes investigating many different allergens.

Therefore, this clinical performance study is conducted to evaluate the diagnostic accuracy of the ALEX² IgE multiplex test using the Multi Array Explorer (MAX 45k, MacroArray Diagnostics) automated laboratory system in comparison to a conventional IgE singleplex test system as well as clinical symptoms and skin prick test results in a total of 826 patients. Patients with the most common inhalant allergies (e.g. grass pollen, house dust mite or cat allergy) will be included as well as patients suffering from Hymenoptera venom allergy, which is the major cause of anaphylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with suspicion of allergy
* Written consent of the participant (and/or his/her parent or legal representative) after being informed

Exclusion Criteria:

* Oral treatment with corticosteroids (>5mg/day)
* Treatment with antihistamines (histamine (H1) receptor blockers)
* Hematological disease (coagulation disorders, anemia)

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy (sensitivity, specificity) of the MAX 45k/ALEX² IgE multiplex test | 1 day
  Sensitivity and specificity of the sIgE status determined by the MAX 45k/ALEX² IgE multiplex test (positive, if ≥0.30 kUA/L) compared to allergy status according to clinical symptoms.

SECONDARY OUTCOMES:
Skin test | 1 day
  Sensitivity and specificity of the sIgE status determined by the MAX 45k/ALEX² IgE multiplex test compared to allergy status according to skin test results (specific for suspected allergy)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Department of Dermatology and Venerology, Medical University of Graz, Graz
  - Allergy Outpatient Clinic Reumannplatz, Vienna

IPD SHARING:
Plan to Share IPD: No